CLINICAL TRIAL: NCT00521690
Title: Safety and Therapeutic Effect of Insulin Detemir in Taiwanese Patients With Type 2 Diabetes Mellitus Not Achieving Glycaemic Targets With OAD With/Without Once-daily NPH Insulin Treatment
Brief Title: The Effect of Insulin Detemir on Blood Glucose Control in Taiwanese Patients With Type 2 Diabetes Failing on OAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1764
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir

SUMMARY:
The trial is conducted in Asia. The aim of the trial is to evaluate the effect of insulin detemir on blood glucose control in Taiwanese patients with type 2 diabetes failing on OAD with/without once-daily NPH Insulin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* HbA1C: 7.0-11.0%
* Previous diabetes treatment for at least 6 months
* BMI max. 35 kg/m2
* Treatment with an oral anti-diabetic drug (OAD)

Exclusion Criteria:

* Type 1 diabetes
* Receipt of any investigational drug within the last three months prior to this trial

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-12; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events, including major hypoglycaemic events | during 16 weeks of insulin detemir therapy

SECONDARY OUTCOMES:
Change in HbA1C | after 16 weeks
Change in weight
Change in fasting plasma glucose (FPG)
Incidence of hypoglycaemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Taipei, Taiwan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com